CLINICAL TRIAL: NCT07046455
Title: Translational Research on the Construction of Trop-2 Targeted PET Probes and Their Application in Advanced Triple-Negative Breast Cancer
Brief Title: Trop-2 Targeted PET Probes in Advanced TNBC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, songguohong, Chief Physician, Deputy Director of the Department, Medical Oncology of Breast Cancer, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Y-Gilead2024-PT-0099
Record Dates: First submitted 2025-06-13; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: TNBC - Triple-Negative Breast Cancer
Keywords: Trop-2; PET probe; triple-negative breast cancer (TNBC)
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET-CT Probe+ Trop-2 ADC (Experimental)
  Interventions: Drug: Sacituzumab Govitecan (SG)

INTERVENTIONS:
Drug: Sacituzumab Govitecan (SG) — After enrollment, before subjects receive TROP-2 ADC treatment, after 2 cycles of treatment, and at the time of progression, in these three phases, subjects will undergo 89Zr-DFO-hSR7 and 18F-FDG examinations once respectively (subjects will first undergo the 18F-FDG examination, and then the 89Zr-DFO-hSR7 examination within 1 week).

SUMMARY:
According to inclusion and exclusion criteria, 20 eligible subjects with triple-negative breast cancer (TNBC) scheduled to receive sacituzumab govitecan were screened. Relevant examination results within 2 weeks before enrollment, including blood and urine routine tests, blood biochemistry, electrocardiogram, serum pregnancy test (for females only), imaging examinations, vital signs, and physical examinations, were collected as baseline assessments to determine whether subjects met enrollment requirements. After enrollment, subjects underwent 89Zr-DFO-hSR7 and 18F-FDG examinations at three time points: before sacituzumab govitecan treatment, after 2 cycles of treatment, and at disease progression. (Subjects first underwent 18F-FDG examination, followed by 89Zr-DFO-hSR7 examination within 1 week.) Within 2 years (with a 1-month window) after completing baseline examinations, investigators will conduct 3-5 follow-ups (at 1 month, 6 months, 1 year, 1.5 years, and 2 years post-examination) via medical record system review or telephone interviews to collect laboratory test results, pathological findings, comprehensive diagnostic results from other imaging modalities, and compare the efficacy of TROP-2 ADC therapy with the results of 89Zr-DFO-hSR7 and 18F-FDG examinations.

This is an exploratory study, initially planned to enroll 20 cases. After obtaining preliminary sample data, further analysis will be conducted to calculate the required sample size. The radiation dose of the drug is approximately 0.02-0.03 mCi/kg. The quality standards for the formulation will be established in accordance with the Chinese Pharmacopoeia (2020 Edition).

DETAILED DESCRIPTION:
1. Primary Objectives To evaluate the correlation between 89Zr-DFO-hSR7 uptake in tumor lesions and TROP2 expression in breast cancer tissues.

   To compare the diagnostic efficacy of 89Zr-DFO-hSR7 and 18F-FDG in breast cancer lesions, including sensitivity, specificity, and accuracy.

   To investigate the validity of 89Zr-DFO-hSR7 in assessing the efficacy of sacituzumab govitecan therapy for breast cancer.
2. Secondary Objectives To clarify the in vivo distribution and metabolism of 89Zr-DFO-hSR7. To monitor resistance to sacituzumab govitecan therapy and explore potential resistance mechanisms.
3. Primary Endpoints The relationship between changes in SUV values on 89Zr-DFO-hSR7 PET imaging before and after sacituzumab govitecan treatment and therapeutic response in breast cancer patients.

   Pathological biopsy results corresponding to suspiciously positive lesions identified by 89Zr-DFO-hSR7 PET imaging.
4. Secondary Endpoints The tumor-to-background ratio (TBR) of standardized uptake values (SUVs) of 89Zr-DFO-hSR7 in target lesions or suspected tumor lesions versus normal tissues within each time window.

To evaluate the in vivo biodistribution of 89Zr-DFO-hSR7 and its temporal changes.

To assess/compare the clinical utility of the probe in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 75 years, male or female, with an ECOG score ≥ 2.
2. Blood routine, liver and kidney functions meet the following standards:

   * Blood routine: Total white blood cell count (WBC) ≥ 3.0×10⁹/L or neutrophil count (Neu) ≥ 1.5×10⁹/L, platelet count (PLT) ≥ 80×10⁹/L, hemoglobin (Hb) ≥ 80 g/L.
   * Liver and kidney functions: Total bilirubin (T - Bil) ≤ 1.5×ULN (upper limit of normal value), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN or ≤ 5×ULN (in case of liver metastasis), serum creatinine (SCr) ≤ 1.5×ULN.
3. Subjects with advanced triple - negative breast cancer previously diagnosed by histopathological diagnosis and imaging evaluation.
4. Expected survival time ≥ 12 weeks.
5. Clinicians assess that TROP - 2 ADC is an appropriate treatment plan for the subject at present.
6. There is at least one measurable target lesion in accordance with the RECIST 1.1 standard.
7. Subjects for whom clinicians recommend PET/CT examination for breast tumor diagnosis and staging.
8. Women of childbearing age (18 - 60 years old) must undergo a pregnancy test within 7 days before the start of the examination and the result is negative; Male and female subjects with fertility must agree to use effective contraceptive measures to ensure no pregnancy during the study period and within 3 months after the examination.
9. The subject can fully understand and voluntarily participate in this experiment, sign the informed consent form, and have good follow - up compliance.

Exclusion Criteria:

1. Severe abnormalities in liver and kidney functions;
2. Women who are in the pre - pregnancy period, pregnant or lactating;
3. Those who cannot lie flat for half an hour;
4. Those who cannot provide informed consent;
5. Those suffering from claustrophobia or other mental illnesses;
6. Those known to be allergic to the investigational drugs or their excipients used in the study treatment;
7. Other situations that the researchers consider make it inappropriate to participate in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
changes in SUV values | Enrollment up for approximately 36 months.
  SUV values of each tumor lesion in 89Zr-DFO-hSR7 PET/CT and 18F-FDG PET/CT imaging before and after sacituzumab govitecan treatment
Pathological biopsy results | Enrollment up for approximately 36 months.
  Pathological biopsy results corresponding to suspiciously positive lesions identified by 89Zr-DFO-hSR7 PET imaging.

SECONDARY OUTCOMES:
The tumor-to-background ratio (TBR) | Enrollment up for approximately 36 months.
  The tumor-to-background ratio (TBR) of standardized uptake values (SUVs) of 89Zr-DFO-hSR7 in target lesions or suspected tumor lesions versus normal tissues within each time window.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided